CLINICAL TRIAL: NCT02170233
Title: SHOCK US STUDY: Fluid Responsiveness in Sepsis Measured by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1406014123
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis: This group will contain patients meeting criteria for sepsis for enrollment in the study (target population).
- Normals: This group will be healthy patients who will have data points recorded for controls for the study to assess the reliability of these measures on healthy patients.

SUMMARY:
The study aim is to examine point-of-care ultrasound findings, reliability, and ease of performance in association with fluid responsiveness for patients with severe sepsis and septic shock. The investigators propose a prospective observational research study of patients presenting to one of three Yale New Haven Hospital emergency departments, York Street Campus, St. Raphael's Campus, and Shoreline Medical Center who meet criteria for sepsis, severe sepsis or septic shock during their emergency department visit.

DETAILED DESCRIPTION:
After each 1 Liter fluid challenge of IV fluid each outcome measure will be repeated to determine if there is a change in ultrasound measures as patients undergo volume resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* All patients age greater than 18 years who meet criteria of sepsis. Septic shock will be defined as those patients with severe sepsis and persistent hypotension (<90mmHg systolic blood pressure) despite a fluid challenge of at least 20cc/kg
* Patients will only be considered eligible for enrollment if the treating physician plans to give at least 1-liter of crystalloid after initial US is performed
* A number (approximately 50 patients) with no symptoms of sepsis will be enrolled to assess measurements in healthy patients. These patients will only have one ultrasound performed for each of the desired study measures.

Exclusion Criteria:

* Patients unable to provide consent such as non-English speaking patients or patient/health care proxy unable to give consent
* History of significant trauma
* Incarcerated patients
* Failure to complete fluid challenge
* Pericardial disease or heart transplant. Patients with left bundle branch block, pulmonary hypertension, known systolic dysfunction (Ejection Fraction <40%), receiving vasopressors, known moderate or severe valvular dysfunction, and irregular heart rhythms will be enrolled but analyzed separately

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to one of three Yale New Haven Hospital emergency departments, York Street Campus, St. Raphael's Campus, and Shoreline Medical Center who meet criteria for severe sepsis or septic shock during their emergency department visit. A number of healthy patients will also be enrolled to act as controls for this study.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness as defined by 15% increase in cardiac output in response to 1 liter of IV fluid | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measurement:
  Carotid corrected flow time in relation to cardiac output to assess fluid responsiveness.

SECONDARY OUTCOMES:
Fluid volume measurement as measured by ultrasound | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measurement:
  IVC diameter in relation to cardiac output to assess fluid responsiveness.
Early (E') septal left ventricular filling velocity as measured by ultrasound | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measurement:
  Early (E') septal left ventricular filling velocity by tissue Doppler in relation to cardiac output to assess fluid responsiveness.
Late (A') septal left ventricular filling velocity as measured by ultrasound | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measure:
  Late (A') septal left ventricular filling velocity by Tissue Doppler in relation to cardiac output to assess fluid responsiveness.
Respirophasic carotid velocity (ΔVpeak) as measured by ultrasound in relation to cardiac output to assess fluid responsiveness. | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measure:
  Respirophasic carotid velocity (ΔVpeak) in relation to cardiac output to assess fluid responsiveness.
Early (E) mitral inflow velocity in relation to cardiac output to assess fluid responsiveness as measured by ultrasound. | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measurement:
  Early (E) mitral inflow velocity in relation to cardiac output to assess fluid responsiveness.
Late (A) mitral inflow velocity in relation to cardiac output to assess fluid responsiveness as measured by ultrasound. | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measurement:
  Late (A) mitral inflow velocity in relation to cardiac output to assess fluid responsiveness.
Carotid velocity-time integral in relation to cardiac output to assess fluid responsiveness as measured by ultrasound. | participants will be followed for the duration of their emergency department stay, an expected average of 6 hours
  Ultrasound Measurement:
  Carotid velocity-time integral in relation to cardiac output to assess fluid responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Moore, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States